CLINICAL TRIAL: NCT07005206
Title: The Effect of Six Hats Thinking Technique on Problem Solving, Critical and Empathic Thinking in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Naciye Esra Koyuncu, Researcher Assistant, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 09.05.2025-E.109769
Record Dates: First submitted 2025-05-14; First posted 2025-06-05 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Nursing Students
Keywords: nursing student; 6 hats thinking; critical thinking; problem solving; empathic thinking

STUDY DESIGN:
Intervention Model Description: This study was conducted as a two-group, experimental design, randomized controlled study.
  Place and Time of the Study The study was conducted with 2nd-year students of the Nursing Department of KTO Karatay University in the spring semester of 2024-2025.
  Population and Sample of the Study The population of the study consisted of all 2nd-year nursing students who were continuing their education and training in the spring semester of 2024-2025. The sample of the study consisted of students who met the inclusion criteria.
  Inclusion Criteria;
  * Taking the Fundamentals of Nursing course
  * Being 18 years of age or older
  * Being able to read and write in Turkish
  * Voluntarily participating in the study Exclusion Criteria;
  * Having taken the Fundamentals of Nursing course before Study termination criteria; Student not participating in two or more case discussions, withdrawing from the study voluntarily.
Who Masked: Participant
Masking Description: Due to the nature of the study, researcher blinding could not be performed. During the statistical analysis phase, the data were transferred to the computer by the researcher and the experimental and control groups were transferred to the SPSS program as '1' and '2', respectively. The statistician was blinded to the groups until all analyses were completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Six Hats Thinking (Experimental): This group received training in the Six Hats Thinking Technique.
  Interventions: Behavioral: Six Hats Thinking; Device: No Intervention (Control)
- classical education (Sham Comparator): This group did not receive any training.
  Interventions: Behavioral: Six Hats Thinking; Device: No Intervention (Control)

INTERVENTIONS:
Behavioral: Six Hats Thinking — A total of 6 sessions of thinking training were given once a week for 6 weeks.
Device: No Intervention (Control) — No intervention was made to this group.

SUMMARY:
This research aims to examine the effect of the Six Thinking Hats Technique application on empathic thinking, critical thinking motivation and problem solving skills in nursing students. In the study, which will be conducted with a pre-test-post-test control group experimental design, the contribution of case discussions made with the Six Thinking Hats Technique to the cognitive and emotional skills of the students will be evaluated.

DETAILED DESCRIPTION:
Nursing education is a dynamic process where theoretical knowledge and clinical practices are integrated; critical thinking, clinical decision-making and problem-solving skills are systematically developed. In this process, in the rapidly changing information society, it is of great importance that nursing students are trained not only as individuals who can access information, but also as professionals who can analyze, interpret information, develop alternative solutions and think in multiple ways. The six thinking hats technique, which aims to develop multi-dimensional thinking skills in nursing students within a systematic structure, is considered an effective teaching method that supports cognitive and emotional development. Within the scope of this technique, it is aimed for individuals to evaluate events and situations in multiple dimensions through six different colored hats, each of which represents a specific way of thinking, such as emotional evaluation, critical thinking, impartial analysis, optimistic perspective, creative thinking and process management.

ELIGIBILITY:
Inclusion Criteria:

* Taking the Fundamentals of Nursing course
* Being 18 years of age or older
* Being able to read and write in Turkish
* Voluntarily participating in the research

Exclusion Criteria:

• Having taken a nursing fundamentals course before

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Problem solving ability | Within 6 weeks after intervention
  Students' problem solving skills will be assessed using the Problem Solving Inventory. Total scores will be compared. The lowest score that can be obtained from the scale is 32, and the highest score is 192.

SECONDARY OUTCOMES:
Critical thinking ability | Within 6 weeks after intervention
  This scale was developed to provide information about motivation for a specific critical thinking task. The scale consists of 19 items, numbered on a Likert-type scale from 1 to 6. Participants are expected to respond by circling the appropriate option for each statement, ranging from 1 to 6 (1 = "Strongly Disagree" and 6 = "Strongly Agree"). These statements express the expectation that each participant will think critically and rigorously (expectation) and the value they place on this type of thinking (value). These statements also include the perceived importance and usefulness of detailed thinking, the sacrifices they will make for this type of thinking, and the interest it generates in them. The scale does not contain reverse items. To score the scale, each question is first assigned a value ranging from 1 to 6. The total score for each subscale is then calculated and divided by the number of items to obtain the mean score. This process is applied separately for the five subscale

OTHER OUTCOMES:
Jefferson Empathy Scale for Nursing Students | Within 6 weeks after intervention
  The original scale consisted of 20 items and three dimensions, while the Turkish version contained 18 items. It was reported that items 5 and 18 in the Turkish version were removed by the researchers because they were found to have low factor loadings. The 18-item Turkish version, like the original, consists of three dimensions. The scale is assessed on a 7-point Likert-type scale ("1 = Strongly Disagree," "2 = Disagree," "3 = Partly Disagree," "4 = Neither Agree nor Disagree," "5 = Partly Agree," "6 = Agree," "7 = Strongly Agree"). Possible scores for the Turkish version range from 18 to 126. Higher scores indicate higher levels of empathy.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to ethical and privacy considerations. Participants did not provide consent for data sharing.